CLINICAL TRIAL: NCT01934036
Title: Efficacy and Safety of Obex®, a Nutritional Supplement, in Overweight or Obese Women
Brief Title: Obex, a Nutritional Supplement, in Overweight and Obese Spanish Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HOPE_TRIAL1
Record Dates: First submitted 2013-08-09; First posted 2013-09-04 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Obesity; Overweight
Keywords: Weight loss; Nutritional supplement; Waist; Body composition; Skinfolds
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Obex, a nutritional supplement (Experimental): Obex will be administered two sachets daily dissolved in a glass of water, 30 minutes before lunch and dinner during two months. Patients will be recommended to comply with a healthy lifestyle through diet and exercise.
  Interventions: Dietary Supplement: Obex
- Placebo (Placebo Comparator): Placebo will be administered two sachets daily dissolved in a glass of water, 30 minutes before lunch and dinner during two months. Patients will be recommended to comply with a healthy lifestyle through diet and exercise.
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Obex — After concluded the two months of treatment, patients will be follow-up during three months without consumption of Obex.
  Arms: Obex, a nutritional supplement
Drug: Placebo — After concluded the two months of treatment, patients will be follow-up during three months without consumption of the placebo.
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the effects of a dietary supplement (Obex®) on anthropometric and physiological variables in Spanish women between 35 and 60 years who are overweight or obese.

DETAILED DESCRIPTION:
The nutritional supplement consists of natural plant extracts such as Caralluma fimbriata, Phaseolus vulgaris, Acai Berry and other antiobesity agents: ornithine, carnitine fumarate, essential fatty acids and certain amino acids, vitamins and minerals.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 35 and 60 years.
* Body Mass Index (BMI) greater than 27 kg/m² and lower than 35 kg/m²
* Ability to provide informed consent

Exclusion Criteria:

* Presence of any endocrine, hepatic, renal or cardiovascular disease.
* History of bariatric surgery
* Pregnancy or lactation
* Concomitant disease with reduced life expectancy
* Severe psychiatric conditions
* Drug dependence

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2013-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of OBEX on skinfolds | Two months of treatment and three months after concluded the treatment
  The primary outcome is to evaluate the effect of the treatment with OBEX on skinfold thickness of the biceps, triceps, subscapular and suprailiac as compared to placebo group at 2 months of treatment.

SECONDARY OUTCOMES:
To evaluate the effect of OBEX on the waist and hip circumferences | Two months of treatment and three months after concluded the treatment
  Waist and Hip circumferences will be measured at baseline and at the end of treatment.
To evaluate the effect of Obex on the arm circumference. | Two months of treatment and three months after concluded the treatment
  The arm circumference will be measured at baseline and at the end of treatment.
To evaluate the effect of Obex on the percentage of body fat | Two months of treatment and three months after concluded the treatment
  Body fat (%) will be assessed at baseline and the end of treatment
To evaluate the effect of Obex on the muscular mass | Two months of treatments and three months after concluded the treatment
  The muscular mass will be measured at baseline and at the end of treatment.
To evaluate the effect of Obex on arterial blood pressures. | Two months of treatment and three months after concluded the treatment
  The arterial BP will be evaluated at baseline and at the end of treatment.
To evaluate the effect of Obex on fasting glucose and cholesterol levels | Two months of treatment and three months after concluded the treatment
  The fasting glucose and cholesterol levels will be evaluated at baseline and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo Prado, Ph.D., Principal Investigator — Universidad Autonónoma de Madrid
Locations (1):
- Universidad Autónoma de Madrid, Ciudad Universitaria de Cantoblanco, Madrid, Spain